CLINICAL TRIAL: NCT02784613
Title: Open-Label Pilot Prospective Vulvoscopy Photography Study of Visible Changes in the Vulva, Vestibule, Vagina Pre/Post 20 Weeks of Daily Administration 60 Mg Ospemifene in Post-Menopausal Women With Dyspareunia From Vulvar Vaginal Atrophy
Brief Title: Vulvoscopy Changes of the Vulva, Vestibule and Vagina With Daily Ospemifene in Women With Dyspareunia From VVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sue Goldstein (Other)
Responsible Party: Sponsor-Investigator, Sue Goldstein, Clinical Research Manager, San Diego Sexual Medicine
Organization: San Diego Sexual Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDSM-2015-02
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Vulvovaginal Atrophy; Dyspareunia
MeSH Terms: conditions — Dyspareunia | interventions — Ospemifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ospemifene open label (Experimental): 60 mg ospemifene daily for 20 weeks
  Interventions: Drug: Ospemifene

INTERVENTIONS:
Drug: Ospemifene — FDA approved medication for the treatment of vulvovaginal atrophy and dyspareunia
  Other Names: Osphena

SUMMARY:
This is an unblinded study to be conducted at a single research center, San Diego Sexual Medicine. Subjects meeting inclusion and exclusion criteria will receive 60 mg ospemifene daily for twenty weeks. After the informed consent is signed, a baseline physical examination, and vulvoscopy with detailed photography of the vulva, vestibule and vagina, will be performed. Physical examination and vulvoscopy with detailed photography of the vulva, vestibule and vagina, will be repeated prospectively every 4 weeks for a total of 20 weeks. Therefore, physical examination and vulvoscopy with detailed photography of the vulva, vestibule and vagina will be performed prospectively at baseline (vulvoscopy session 1), 4 weeks (vulvoscopy session 2), 8 weeks (vulvoscopy session 3), 12, weeks (vulvoscopy session 4), 16 weeks (vulvoscopy session 5) and 20 weeks (vulvoscopy session 6) following daily administration of 60 mg ospemifene.

DETAILED DESCRIPTION:
Ospemifene is indicated for post-menopausal women diagnosed with vulvar vaginal atrophy (VVA) and dyspareunia. While ospemifene clinically significantly reduces pain associated with dyspareunia, there has been little prospective documentation using vulvoscopy with detailed photography of the visible changes to the vulva, vestibule and vaginal region with daily administration of 60 mg ospemifene in post-menopausal women with VVA and dyspareunia. This study will include a total of 6 prospective photographic sessions of the vulva, vestibule and vagina over the 20 weeks administration of 60 mg ospemifene in the study. Comparisons will be made of baseline photography (vulvoscopy session 0) with photography at 4 weeks (vulvoscopy session 1), 8 weeks (vulvoscopy session 2), 12 weeks (vulvoscopy session 3), 16 weeks (vulvoscopy session 4) and 20 weeks (vulvoscopy session 5).

Currently there have been limited prospective studies using vulvoscopy with detailed photography demonstrating visible changes to the vulva, vestibule and vagina following oral administration of 60 mg ospemifene in post-menopausal women with VVA and dyspareunia. Information regarding visible changes to the vulva, vestibule and vagina may be very important to the patient and to the health care provider to best understand the beneficial effects of ospemifene and to ensure patient compliance with treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent and HIPAA authorization before any study procedures are conducted
2. Subject is female
3. Subject is aged 21-80 years
4. Subject has a body mass index (BMI) < 37 kg/m2
5. Subject is menopausal either naturally (at least 12 months amenorrheic) or 6 weeks after a bilateral salpingo-oophorectomy prior to natural menopause subjects with hysterectomy only must have a serum Follicle Stimulating Hormone > 40 milli-International unit /mL
6. Subject has vulvovaginal atrophy with dyspareunia
7. Subject has had a normal mammogram within the last 6 months
8. Subject has normal pap smear within last 6 months
9. Subject has an endometrial stripe ≤ 4 mm within the last 6 months if she has a uterus
10. Subject agrees to comply with the study procedures and visits.

Exclusion Criteria:

1. Subject has a hypersensitivity to any of the ingredients of ospemifene
2. Subject has used ospemifene in the past
3. Subject has documented or suspected breast cancer, history of heart attack or stroke
4. Subject has clinically significant findings on physical examination
5. Subject has uncontrolled hypertension
6. Subject has any chronic medical condition or psychologic disorder that the Principal Investigator feels makes her ineligible for the study
7. Subject is currently on local or systemic androgen therapy including local or systemic testosterone (washout 14 days for local or topical androgen or non-depot injection, 1 month for depot, 6 months for pellet
8. Subject is currently on local or systemic estrogen therapy or androgen therapy (washout 14 days for vaginal estrogen, 60 days for oral/transdermal therapy)
9. Subject is currently using a Selective Estrogen Receptor Modulator (SERM) or products that have estrogenic or anti-estrogenic effects within last month
10. Subject currently using itraconazole, ketoconazole, digitalis or alkaloids heparin or strong cytochrome P 450 3A4 inhibitors
11. Subject has a history of substance abuse within 12 months prior, or consuming > 14 alcoholic drinks per week
12. Subject has received an investigational drug within 30 days prior to signing consent
13. Subject has any condition or exhibits behavior that indicates to the Principal Investigator that the Subject is unlikely to be compliant with study procedures and visits.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2017-02-07 (Actual); Study Completion 2017-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Goldstein, MD, Principal Investigator — San Diego Sexual Medicine
Locations (1):
- San Diego Sexual Medicine, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Information will be combined and not reported as individual participant data.

REFERENCES:
- [Background] Bachmann GA, Komi JO; Ospemifene Study Group. Ospemifene effectively treats vulvovaginal atrophy in postmenopausal women: results from a pivotal phase 3 study. Menopause. 2010 May-Jun;17(3):480-6. doi: 10.1097/gme.0b013e3181c1ac01. PMID 20032798
- [Background] Portman DJ, Bachmann GA, Simon JA; Ospemifene Study Group. Ospemifene, a novel selective estrogen receptor modulator for treating dyspareunia associated with postmenopausal vulvar and vaginal atrophy. Menopause. 2013 Jun;20(6):623-30. doi: 10.1097/gme.0b013e318279ba64. PMID 23361170
- [Background] Goldstein SR, Bachmann GA, Koninckx PR, Lin VH, Portman DJ, Ylikorkala O; Ospemifene Study Group. Ospemifene 12-month safety and efficacy in postmenopausal women with vulvar and vaginal atrophy. Climacteric. 2014 Apr;17(2):173-82. doi: 10.3109/13697137.2013.834493. Epub 2013 Nov 23. PMID 23984673
- [Background] Simon JA, Lin VH, Radovich C, Bachmann GA; Ospemifene Study Group. One-year long-term safety extension study of ospemifene for the treatment of vulvar and vaginal atrophy in postmenopausal women with a uterus. Menopause. 2013 Apr;20(4):418-27. doi: 10.1097/gme.0b013e31826d36ba. PMID 23096251
- [Result] Goldstein SW, Winter AG, Goldstein I. Improvements to the Vulva, Vestibule, Urethral Meatus, and Vagina in Women Treated With Ospemifene for Moderate to Severe Dyspareunia: A Prospective Vulvoscopic Pilot Study. Sex Med. 2018 Jun;6(2):154-161. doi: 10.1016/j.esxm.2018.03.002. Epub 2018 Apr 18. PMID 29678557

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ospemifene Open Label
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Baseline assessments made for completers only
Arm/Group | Ospemifene Open Label
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Visible Changes to the Vulva, Vestibule and Vaginal Region on Photography
Description: Change in score on the Vulvoscopic Genital Tissue Appearance (VGTA) scale from baseline to 20 weeks was measured using ten parameters: 1) loss of labia majora, 2) loss of labia minora, 3) decreased glans clitoris, 4) prominence of the urethral meatus, 5) stenosis of the introitus, 6) vestibular pallor, 7) vestibular erythema, 8) loss of vestibular moisture, 9) loss of vaginal rugae, and 10) loss of prominence of the anterior vaginal wall to determine health of the vulva, vestibule and vaginal region using vulvoscopic photographs. VGTA scoring ranges from 0 (normal) to 3 (most severe) for each parameter, for a total score ranging from 0 (normal) to 30 (most severe). Each region assessed is reflected as worse for a higher score and better for a lower score in the 0-3 range, and the same for the total score, with 0 being the best possible score and 30 the worse.
Time Frame: Baseline and 20 weeks
Measure: Median (Inter-Quartile Range); unit: points improvement on VGTA scale
Groups:
- Open Label: 60 mg ospemifene daily for 20 weeks
  Ospemifene: FDA approved medication for the treatment of vulvovaginal atrophy and dyspareunia
Arm/Group | Open Label
Number analyzed (Participants) | 8
points improvement on VGTA scale | 8 [7 to 8]
Statistical Analysis 1: Comparison: Open Label; Test type: Superiority; p = 0.05, t-test, 2 sided — Differences in pre- and post-treatment scores were compared using Wilcoxon signed-rank test for non-parametric matched pairs. All tests of significance were 2-tailed. All analyses were performed in Stata®, version 13

2. Secondary Outcome: Changes in Pain Scale
Description: Changes in pain as noted on the pain scale (0-3) by q-tip testing of the vestibule by the clinician, with 0 representing no pain at the location and 3 being severe in each location, 1 o'clock, 3 o'clock, 5 o'clock, 6 o'clock, 7 o'clock, 9 o'clock and 11 o'clock circling the vestibule. The maximum total pain score range is 0 (no pain) to the worst score possible of 21 indicating severe pain at all locations.
Time Frame: Baseline and 20 weeks
Population: Completers
Measure: Median (Inter-Quartile Range); unit: points improvement
Arm/Group | Open Label
Number analyzed (Participants) | 8
points improvement | 10 [9.5 to 13]

3. Secondary Outcome: Percentage of Sexual Encounters in Which Pain Was Experienced
Description: For each sexual encounter, patients were required to record a ''yes" or "no" response to the following question: Did you experience pain during intercourse? The percentage of sexual encounters in which the woman answered "yes" to this question at baseline (first month of the study) and at week 20 (last month of the study) was compared. The worst score possible was experiencing pain during 100% of sexual encounters and the best possible score was experiencing pain during 0% of sexual encounters at any given assessment period.
Time Frame: Baseline and 20 weeks
Population: completers
Measure: Median (Inter-Quartile Range); unit: percentage of sexual encounters
Arm/Group | Open Label
Number analyzed (Participants) | 8
percentage of sexual encounters
  Baseline value | 80 [20 to 100]
  Week 20 value | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 6 months per participant
Description: clinical trials dot gov definitions used
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=8)
microscopic hematuria (Renal and urinary disorders) | 1 (1) — Noted in urine at end of study but no urine sample taken at screening for comparison
influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sinus infection (Infections and infestations) | 1 (1) — medication from sinus infection caused diarrhea for participant
diarrhea (Gastrointestinal disorders) | 1 (1) — Caused by medication from sinus infection
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — during acute coryza
acute coryza (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small pilot study size; open label without placebo; reader of vulvoscopic photographs was not involved in any part of data collection or subject visits but was aware of whether the photos were from baseline or end of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT02784613/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT02784613/SAP_001.pdf
  • Informed Consent Form (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT02784613/ICF_002.pdf